CLINICAL TRIAL: NCT06764433
Title: Efficacy of Greater Occipital Nerve Pulsed Radiofrequency Treatment At C2 Level in Cervicogenic Headache
Brief Title: Greater Occipital Nerve Pulsed Radiofrequency in Cervicogenic Headache
Acronym: GONPRF CEH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ülkü Sabuncu, assoc prof dr, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1-23-3686; turkısh health ministry (Other: Bilkent Ankara City Hospital)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Headache, Cervicogenic; Cervicogenic Headache
Keywords: Cervicogenic headache, proximal GON PRF, Ultrasound guided, C2 level
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, comparative, observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical data of the patients before and after treatment will be compared (Other): According to the International Classification of Headache Disorders (ICHD)-III diagnostic criteria, patients diagnosed with cervicogenic headache will undergo a proximal technique C2 level greater occipital nerve (GON) diagnostic block under ultrasound (USG) guidance, and patients with a positive response (≥50% reduction in pain or positive effect) will receive GON-PRF treatment with the same technique.
  This study mainly aims to evaluate the clinical efficacy and safety of GON PRF treatment applied at the C2 level under USG guidance in cervicogenic headache during the follow-up period.
  Our secondary aim is to determine the effects of the GON PRF treatment we applied on the analgesic drug consumption, daily life activities and sleep of the volunteers, how they generally perceive this treatment and whether there is a need for any additional treatment.
  Interventions: Procedure: GONPRF; Procedure: Proximal GONPRF

INTERVENTIONS:
Procedure: GONPRF — GON PRF treatment, which we apply by imaging the target nerve and surrounding structures with the proximal technique (at C2 level) under USG guidance in patients who do not respond to conservative treatments for cervicogenic headache.
Procedure: Proximal GONPRF — Ultrasound-guided pulsed radiofrequency treatment of the greater occipital nerve at the C2 level

SUMMARY:
The effect of GON PRF treatment applied with USG-guided proximal technique in patients who do not respond to conservative treatments for cervicogenic headache

DETAILED DESCRIPTION:
In our study, GON PRF will be applied to volunteers who are diagnosed with cervicogenic headache according to ICHD-3 criteria, who meet the study criteria and who report a positive effect with diagnostic GON block application. The main purpose of our study is to evaluate the clinical efficacy and safety of ultrasound-guided C2 level greater occipital nerve pulsed radiofrequency treatment in cervicogenic headache during the follow-up period. Our secondary purpose is to determine the effects of the GON PRF treatment we applied on the volunteers' analgesic drug consumption, daily life activities and sleep, how they generally perceive this treatment and whether there is a need for any additional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervicogenic headache according to ICHD-3 criteria
* Cranial and cervical spine imaging is available
* Number of headache days per month 5 and/or more
* Inadequate benefit from pharmacological treatments or physical therapy methods used
* Volunteer patients who can understand and approve the treatment and the informed consent form and who can comply with the treatment

Exclusion Criteria:

* History of secondary headache other than cervicogenic headache according to ICHD-3 criteria
* Cervical nerve root irritation and/or spinal stenosis symptoms and signs
* Sensory deficit findings in the greater occipital nerve dermatome
* Craniocervical defect or other anatomical abnormality in the target area or nearby the procedure
* Local or systemic infection
* Received nonpharmacological treatment within the last 3 months (physical therapy, botulinum toxin A, acupuncture, ozone, cognitive behavioral therapy, etc.)
* Pregnancy or suspected pregnancy
* Known allergy to local anesthetic drugs
* History of malignancy
* Known organic disease of the brain and spinal cord
* History of cranial/cervical surgery within the last 1 year
* Bleeding-clotting disorder or oral anticoagulant use
* Comorbid disease that may cause headache (uncontrolled hypertension, intracranial lesion, etc.)
* Compliance with treatment and treatment results diseases that may affect the evaluation (psychiatric disorder, dementia, etc.)
* Those who request re-treatment due to the emergence of contralateral pain or other types of pain during the follow-up period after treatment
* Those who do not accept treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 3 months
  Average headache severity, maximum headache severity, number of headache days (monthly) measured with a visual analog scale (VAS; 10-point VAS scoring, 0 being no pain and 10 being the highest pain intensity that can be tolerated)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I dont want to.

REFERENCES:
- [Background] Gabrhelik T, Michalek P, Adamus M. Pulsed radiofrequency therapy versus greater occipital nerve block in the management of refractory cervicogenic headache - a pilot study. Prague Med Rep. 2011;112(4):279-87. PMID 22142523
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31337167/